CLINICAL TRIAL: NCT02757248
Title: A Phase I Trial of Volasertib Plus Romidepsin in Patients With Relapsed/Refractory Peripheral T Cell and Cutaneous T Cell Lymphoma
Brief Title: Ph1 Volasertib Plus Romidepsin in R/R PTCL and CTCL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Boehringer Ingelheim is discontinuing their volasertib development program
Sponsor: Anne Beaven, MD (Other)
Collaborators: National Comprehensive Cancer Network (Network); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Anne Beaven, MD, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00060068
Record Dates: First submitted 2016-03-22; First posted 2016-05-02 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: PTCL; CTCL
MeSH Terms: interventions — BI 6727; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Volasertib 75mg/m2 on days 1 and 8 Romidepsin 12mg/m2 on days 1, 8 and 15
  Interventions: Drug: Volasertib; Drug: Romidepsin
- Cohort 2 (Experimental): Volasertib 100mg/m2 on days 1 and 8 Romidepsin 12mg/m2 on days 1, 8 and 15
  Interventions: Drug: Volasertib; Drug: Romidepsin
- Cohort 3 (Experimental): Volasertib 100mg/m2 on days 1 and 8 Romidepsin 14mg/m2 on days 1, 8 and 15
  Interventions: Drug: Volasertib; Drug: Romidepsin
- Cohort 4 (Experimental): Volasertib 150mg/m2 on days 1 and 8 Romidepsin 14mg/m2 on days 1, 8 and 15
  Interventions: Drug: Volasertib; Drug: Romidepsin
- Cohort -1 (Experimental): Volasertib 50mg/m2 on days 1 and 8 Romidepsin 10mg/m2 on days 1, 8 and 15
  Interventions: Drug: Volasertib; Drug: Romidepsin

INTERVENTIONS:
Drug: Volasertib — Volasertib 75-150mg/m2 given intravenously on days 1 and 8
Drug: Romidepsin — Romidepsin 12-14mg/m2 given intravenously on days 1, 8 and 15

SUMMARY:
This is a phase I study of the combination of volasertib and romidepsin in patients with relapsed/refractory peripheral T cell lymphoma (PTCL) or stage IIB-IV cutaneous T cell lymphoma (CTCL). This study will determine the maximum tolerated dose (MTD) of this combination by treating cohorts of patients at a certain dose combination. The investigators will use a Bayesian design to determine the dose combination for the next cohort of patients and to determine the MTD. Overall response rate as well as adverse events will be monitored and reported.

DETAILED DESCRIPTION:
This is a non-randomized, unblinded single arm Phase I multi-center trial to determine the maximum tolerated dose (MTD) of the combination of volasertib and romidepsin in patients with relapsed/refractory peripheral T cell (PTCL) and cutaneous T cell (CTCL) lymphoma.

Primary Objectives:

1. Determine the maximum tolerated dose (MTD) of the combination of romidepsin and volasertib in patients with relapsed/refractory peripheral T cell and cutaneous T cell lymphoma.

Secondary Objectives:

1. Evaluate the overall response rate (ORR) to the combination of romidepsin and volasertib in patients with relapsed/refractory peripheral T cell and cutaneous t cell lymphoma.
2. Define gene expression signatures and patterns of acquired tumor mutations that dynamically correlate to clinical response to romidepsin/volasertib combination therapy in cutaneous T cell lymphoma (CTCL) through longitudinal RNA sequencing of tumor samples.

Dose Combinations

(-1): Volasertib 50mg/m2 Days 1 & 8; Romidepsin 10mg/m2 Days 1, 8 & 15

(1-starting dose): Volasertib 75mg/m2 Days 1 & 8; Romidepsin 12mg/m2 Days 1, 8 & 15 (2): Volasertib 100mg/m2 Days 1 & 8; Romidepsin 12mg/m2 Days 1, 8 and 15 (3): Volasertib 100mg/m2 Days 1 & 8; Romidepsin 14mg/m2 Days 1, 8 and 15 (4): Volasertib 150mg/m2 Days 1 & 8; Romidepsin 14mg/m2 Days 1, 8 and 15

Each cycle is 28 days Each drug is given intravenously

ELIGIBILITY:
Inclusion Criteria:

1. A) Patients with a relapsed/refractory peripheral T cell lymphoma. Patients must have received at least one prior standard cytotoxic regimen such as CHOP or EPOCH OR B) Patients with relapsed/refractory stage IIb-IV cutaneous T cell lymphoma who have received at least one standard systemic treatment such as extracorporeal photopheresis, bexarotene or interferon.
2. Age > 18 years old
3. Eastern Cooperative Oncology Group performance status of <2
4. Evidence of measurable or evaluable disease
5. Patients must have recovered from all clinically relevant toxicities related to prior anticancer therapies to ≤ grade 2 (CTCAE v 4.03). Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.
6. Platelets >100 x 109/L
7. ANC>1.5 x 109/L
8. AST/ALT <3.0 x institutional ULN, except for people with liver involvement by their lymphoma, who may be included if AST/ALT <5 x ULN.
9. Total Bilirubin < 1.5 x ULN, except for patients with gilbert's syndrome who may be included if total bilirubin < 3.0 x ULN and direct bilirubin < 1.5 x ULN
10. The following laboratory values must be greater than the lower limits of normal prior to starting study drug (supplementation allowed): potassium, magnesium
11. Calculated or measured CrCl> 30ml/min (Appendix: 3)
12. Ability to provide written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
13. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Prior Treatment:

   1. Patients must not have received chemotherapy, radiation or surgical resection of malignancy within 3 weeks prior to the start of study drug. However, if they have received nitrosurea or mitomycin C then they should not be enrolled in the study until 6 weeks after therapy was last received.
   2. No limitations to number of prior therapies.
   3. Prior treatment with volasertib or any PLK1 inhibitor
   4. Prior treatment with a histone deacetylase inhibitor (anti-epileptics ok)
2. Active, uncontrolled, serious infection or medical or psychiatric illness likely to interfere with participation in this clinic trial
3. Known HIV infection.
4. Active or chronic hepatitis B infection.
5. Clinical evidence of symptomatic progressive brain or leptomeningeal disease during the past 6 months.
6. Pregnant or breast feeding. Treatment under this protocol would expose an unborn child to significant risks.
7. Women and men of reproductive potential who are unwilling or unable to use an effective means of birth control during the study and for 3 months after receiving study drug.
8. Major surgery within the four weeks prior to initiating protocol therapy.
9. Diagnosis or treatment for any malignancy other than NHL within the 3 years preceding Day 1 of the protocol therapy. Exceptions are:

   1. Basal or squamous cell carcinoma of the skin
   2. In situ malignancy that has been completely resected.
   3. Prostate cancer that was treated with prostatectomy or radiotherapy over 2 years before Day 1 of protocol therapy and whose PSA is undetectable.
10. Treatment with another investigational agent currently or within 21 days prior to enrollment. Patients may participate in other non-treatment studies concurrently if it will not interfere with participation in this study.
11. Myocardial infarction or unstable angina within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
12. QTcF>470msec using the Fredericia formula.
13. Known hypersensitivity to the trial drugs (volasertib and romidepsin)
14. Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with study drug and for the duration of participation (see Appendix 2 Tables):

    1. Medication with a significant known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
    2. Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    3. Herbal supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months or until 2 DLTs are experienced in a cohort
  Determine the maximum tolerated dose (MTD) of the combination of romidepsin and volasertib in patients with relapsed/refractory peripheral T cell and cutaneous T cell lymphoma.

SECONDARY OUTCOMES:
Overall Response Rate | 24 months
  Evaluate the overall response rate (ORR) to the combination of romidepsin and volasertib in patients with relapsed/refractory peripheral T cell and cutaneous t cell lymphoma.
Gene Expression Signature | 60 months
  Define 1) genes expressed at significantly different levels (using linear analysis or the Wilxocon rank sum test and p< 0.05 as significance threshold) in tumor biopsies taken before treatment from patients exhibiting a clinical response versus non-responders to romidepsin/volasertib by analysis of levels of mRNA gene transcription by mRNA whole transcriptome sequencing (RNA-seq) Comparison of baseline to interim 8 week biopsy samples will be used to define changes in gene expression induced by combination treatment. These will be derived for each patient by using paired T tests for RNA sequencing FPKM values with correction for multiple comparisons via FDR calculation by the Benjamini-Hochberg method (a cutoff of FDR < 0.05 will be used to define genes included in the treatment gene signature).
Gene Mutation Analysis | 60 months
  Define 2) and 2) define mutations associated with primary (lack of clinical response) or acquired resistance (relapse or loss of response after first clinical response) to romidepsin/volasertib by analysis of tumor genetic sequences by using RNA-seq metholodies on tumor samples taken before or after treatment with romidepsin/volasertib and analysis of paired normal DNA sequence(s). Mutations for relapse samples will be obtained by comparing transcriptome profiles before and after development of resistance to romidepsin/volasertib. Specifically, we will assess whether individual genes become mutated at relapsed in a recurrent fashion (in 2 or more patients in the cohort).

CONTACTS AND LOCATIONS:
Overall Officials: Anne w Beaven, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No